CLINICAL TRIAL: NCT02141529
Title: Bipolar Versus Unipolar Intraarticular Pulsed Radiofrequency Thermocoagulation in Chronic Knee Pain Treatment: A Prospective Randomized Study
Brief Title: Intraarticular Pulse Radiofrequency to Treat Chronic Knee Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Ersel GULEC, Assist.Prof., Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IAPRF01
Record Dates: First submitted 2014-05-15; First posted 2014-05-19 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Osteoarthritis
Keywords: Intraarticular; pulsed radiofrequency; osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Unipolar PRF (Active Comparator): Unipolar pulsed radiofrequency thermocoagulation, intraarticularly in knee joint, 42oC of temperature during ten minutes
  Interventions: Procedure: Unipolar pulsed radiofrequency thermocoagulation
- Bipolar PRF (Experimental): Bipolar pulsed radiofrequency thermocoagulation, intraarticularly in knee joint, 42oC of temperature during ten minutes
  Interventions: Procedure: Bipolar pulsed radiofrequency thermocoagulation

INTERVENTIONS:
Procedure: Unipolar pulsed radiofrequency thermocoagulation — Unipolar pulsed radiofrequency thermocoagulation, intraarticular administration into the knee joint
  Arms: Unipolar PRF
Procedure: Bipolar pulsed radiofrequency thermocoagulation — Bipolar pulsed radiofrequency thermocoagulation, intraarticular administration into the knee joint
  Arms: Bipolar PRF

SUMMARY:
The purpose of this study is to determine whether bipolar intraarticular pulsed radiofrequency method has a superiority to unipolar mode in the treatment of chronic knee pain.

DETAILED DESCRIPTION:
After obtaining written informed consent and ethics committee approval, 100 patients aged 20-70 years with osteoarthritis having knee pain over 3 months are recruited to the randomized, double-blind study. Exclusion criteria are a chronic knee pain caused by infection, inflammation, tumors, and fractures or a history of acute knee pain, previous knee surgery, connective tissue diseases, neurologic or psychiatric disorders, administration of steroids or hyaluronic acids within the last three months, coagulation disorders and local infection at the site of intervention planned.

Patients are admitted to the preoperative unit 15 minutes before the procedure. After intravenous access is established by a 20 gauge cannula, all patients are monitored with non-invasive blood pressure (NIBP), electrocardiogram (ECG) and peripheral oxygen saturation (SpO2) (Drager-Primus Anesthesia Device Monitor, Drager Medical Systems, Inc 16 Electronics Avenue, Denver, MA 01923 USA) in the operating room before the beginning of procedure. Patients are randomly allocated into two groups in a 1:1 ratio by a computer-generated list. Allocation is provided with sealed envelopes containing group named paper.

After patients are positioned to supine, a pillow is placed to support below their knee to be treated. Anteroposterior (AP) fluoroscopic image of the knee joint is obtained with C-arm fluoroscopy. 1% of lidocaine is injected 2 ml under the skin at locations corresponding to joint space both of sides of the patellar ligament and A 10 cm 22-gauge two radiofrequency electrode needles with a 5 mm active tip (NeuroTherm® RF Cannula) are bilaterally inserted at the same points and advanced under fluoroscopic guidance entering the cavity of the knee joint at the both medial and lateral sites until needle tips are in the middle of the joint space. Pulsed Radiofrequency (PRF) is bilaterally performed in 42oC of temperature during ten minutes. After positioned to supine, a pillow is placed to support below their knee at the planned procedure site. Anteroposterior (AP) fluoroscopic image of the knee joint is obtained with C-arm fluoroscopy. Under fluoroscopy at locations corresponding to joint space both of sides of the patellar ligament, 1% of lidocaine is injected 2 ml under the skin and at the same points with 22 gauge of thickness, 10 cm in length, 5 mm of length active tipped two radiofrequency electrode needles (NeuroTherm® RF Cannula) are bilaterally inserted and advanced under fluoroscopy entering the cavity of the knee joint at the both medial and lateral sites until needle tips are in the middle of the joint space. PRF is bilaterally performed with a unipolar mode, 45V voltage, 2 Hz frequency, at a temperature of 42oC, 10 msec pulse width for 10 minutes in group U. The same procedure is bilaterally performed with a bipolar mode for 10 minutes in group B. All procedures are performed by one practitioner who is not informed about the type of procedure (unipolar or bipolar mode) and also patients are not aware of which type of treatment received.

If any complication is not observed for one hour after the procedure, the patients are discharged. Paracetamol is prescribed for the supplemental analgesic requirement.

The degree of pain is assessed with a 10-cm VAS. "0" identifies the least possible pain and "10" determines the most severe pain that can be considered. We evaluate the health status of patients by the WOMAC index which is valid and reliable self-administered questionnaire including 24 items divided into 3 subscales (pain, stiffness, and physical function).(1,2) Visual Analog Scale (VAS) and Western Ontario and McMaster Universities Osteoarthritis Index LK 3.1 (WOMAC) and supplemental analgesic requirements, any side effects and complications such as a motor or sensorial loss are recorded in both groups at before the procedure and at 1, 4, and 12 weeks after the procedure. We assess the patients when they are requested to our clinic for clinical examination. We also call them by telephone to any further advice.

The primary outcomes are VAS scores measuring knee pain at 1, 4, and 12 weeks after the procedure. Secondary outcomes are WOMAC scores to evaluate the quality of life and the functional response of treatment of patients and the incidence of adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 20-70 years
* Patients with osteoarthritis having knee pain over 3 months

Exclusion Criteria:

* Chronic knee pain caused by infection, inflammation, tumors, and fractures
* A history of acute knee pain, previous knee surgery, connective tissue diseases, neurologic or psychiatric disorders,
* The administration of steroids or hyaluronic acids within the last three months
* Coagulation disorders
* Local infection at the site of intervention planned

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-05; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale scores to measure the pain degree | 12 weeks

SECONDARY OUTCOMES:
WOMAC scores to measure the degree of quality of life and the functional response of treatment of patients | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ersel Gulec, Assist.Prof., Principal Investigator — Cukurova University Faculty of Medicine
Locations (1):
- Cukurova University Faculty of Medicine Research Hospital, Adana, Turkey (Türkiye)

REFERENCES:
- [Result] Bellamy N, Buchanan WW, Goldsmith CH, Campbell J, Stitt LW. Validation study of WOMAC: a health status instrument for measuring clinically important patient relevant outcomes to antirheumatic drug therapy in patients with osteoarthritis of the hip or knee. J Rheumatol. 1988 Dec;15(12):1833-40. PMID 3068365
- [Result] Tuzun EH, Eker L, Aytar A, Daskapan A, Bayramoglu M. Acceptability, reliability, validity and responsiveness of the Turkish version of WOMAC osteoarthritis index. Osteoarthritis Cartilage. 2005 Jan;13(1):28-33. doi: 10.1016/j.joca.2004.10.010. PMID 15639634
- [Result] Choi WJ, Hwang SJ, Song JG, Leem JG, Kang YU, Park PH, Shin JW. Radiofrequency treatment relieves chronic knee osteoarthritis pain: a double-blind randomized controlled trial. Pain. 2011 Mar;152(3):481-487. doi: 10.1016/j.pain.2010.09.029. Epub 2010 Nov 4. PMID 21055873
- [Result] Sluijter ME, Teixeira A, Serra V, Balogh S, Schianchi P. Intra-articular application of pulsed radiofrequency for arthrogenic pain--report of six cases. Pain Pract. 2008 Jan-Feb;8(1):57-61. doi: 10.1111/j.1533-2500.2007.00172.x. No abstract available. PMID 18211593
- [Derived] Gulec E, Ozbek H, Pektas S, Isik G. Bipolar Versus Unipolar Intraarticular Pulsed Radiofrequency Thermocoagulation in Chronic Knee Pain Treatment: A Prospective Randomized Trial. Pain Physician. 2017 Mar;20(3):197-206. PMID 28339432